CLINICAL TRIAL: NCT03803722
Title: A Prospective Multicenter, Comparative, Randomized, Single-blind, Non-inferiority Study of Eyestil Protection® Unidose Versus Vismed® Unidose in Patients With Moderate to Severe Dry Eye Syndrome
Brief Title: To Demonstrate the Non-inferiority of Eyestil Protection® Compared to Vismed® in Terms of Clinical Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment process and COVID situation worsened the situation. SIFI has developed a new product with probably a better performance. SIFI changed its marketing strategy and decided that Eyestil® Protection will be not marketed anymore
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 048/SI
Record Dates: First submitted 2018-12-10; First posted 2019-01-15 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Approximately 80 patients globally: 40 per arm with a 1:1 ratio including an expected dropout rate of 15%. Single masked. Medical Device
Who Masked: Investigator
Masking Description: Single Blind: investigator masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A Eyestil Protection® (Experimental): No inferiority of Eyestil Protection® unidose versus Vismed® unidose The intervention consists of Eyestil Protection® : sterile preservative free, medical device, class IIa and CE marked. It contains 0.2% xanthan gum, presented in 0.3 ml unidose containers. It is not available yet on the French Market.
  dosage: 6 drops a day for three months period.
  Interventions: Device: Eyestil Protection® unidose
- Arm B Vismed® (No Intervention): Vismed®: sterile preservative free, medical device class IIb and CE marked. It contains 0.18% sodium hyaluronate, presented in 0.3 ml unidose containers. It is already on the French market.
  dosage: 6 drops a day for three months period.

INTERVENTIONS:
Device: Eyestil Protection® unidose — to demonstrate the non-inferiority of Eyestil Protection® in terms of performance and safety, when compared to Vismed® in treatment of dry eye disease.
  Arms: Arm A Eyestil Protection®

SUMMARY:
This is a national, prospective, multicenter, comparative, randomized, single-blinded non-inferiority study performed in two parallel groups.

3 months (plus a run in period of 15 days prior inclusion) Patients with moderate to severe dry eye syndrome.

DETAILED DESCRIPTION:
Public hospitals and private practices specialized in ophthalmology Approximately 10 sites France Approximately 80 patients globally: 40 per arm with a 1:1 ratio including an expected dropout rate of 15%.

Dry eye has been defined as a multifactorial disease of the ocular surface characterized by a loss of homeostasis of the tear film and accompanied by ocular symptoms, in which the tear film instability and hyperosmolarity, ocular surface inflammation and damage, and neurosensory abnormalities play etiological roles.

However, prevalence estimates for dry eye vary dramatically from 5% to 50% due to the various operational definitions of dry eye used and the characteristics of the population studied.

The available evidence suggests also that dry eye has a negative impact on overall quality of life. It causes pain and irritation and affects ocular and general health and well-being, the perception of visual function and visual performance. Reduced quality of life in everyday activities and leisure pursuits is reported by 60% of patients, while 38% of patients complain of reduced efficiency at work.

Therefore, the economic burden and impact of dry eye on vision and quality of life, work productivity, psychological and physical impact of pain are considerable. As a consequence, dry eye represents a public health burden. However, only a handful of therapies are available for dry eye patient and are used according to the disease severity.

In such context, SIFI SpA. has developed Eyestil Protection® (or SF-104 XNT Single dose). It is a sterile preservative-free device (eye drops) for ophthalmic use containing 0.2% xanthan gum, presented in 0.3 ml unidose containers. The main action of Eyestil Protection is to lubricate and moisturize the ocular surface as well as to protect it from oxidative stress thanks to the anti-oxidative properties of the xanthan gum (as demonstrated by in-vitro studies (Amico, Tornetta et al. 2015). It is indicated in all cases of dry-eye related ocular discomfort and to relief ocular discomfort due to the use of contact lenses.

Eyestil Protection® unidose is CE marked but is not available yet in all European countries, notably in France.

Confronted to a European regulatory change on medical devices - from a Directive (Directive 1993/42/EEC) to a Regulation (MDR 2017/745) that now requires clinical evidence of device performance and safety; SIFI SpA decided to implement the present clinical comparative performance study. The choice of Vismed® (unidose) as the comparator has been done since it is the current French standard of care treatment for patients with moderate to severe dry eyes.

Primary objective

• To demonstrate the non-inferiority of Eyestil Protection® compared to Vismed® in terms of clinical performance as detected by a reduction of keratitis lesions objectified by staining tests after 1 month of treatment, in patients with moderate to severe dry eye syndrome with keratoconjunctivitis.

Secondary objectives Clinical performance

* To evaluate the tear film stability per group as objectified by the tear break up time (TBUT) test at month 1 and 3;
* To evaluate the long term clinical performance of Eyestil Protection® compared to Vismed® as detected by a reduction of keratitis lesions objectified by staining tests after 3 months of treatment;
* To evaluate the tear production per group as objectified by the Schirmer test at month 3.

Patient reported outcomes

* To compare patients reported outcomes (PRO) measures per group at month 1 and 3, including:

  * Patient's reported symptoms and
  * Patient's quality of life (QoL). Investigator overall satisfaction
* To assess investigator's overall satisfaction of the treatment's clinical performance at month 1 and 3.

Safety • To describe the safety profile of Eyestil Protection® compared to Vismed® after 3 months of treatment.

Exploratory objectives

• To compare patient's QoL subscale scores per group at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, male or female, of at least 18 years of age at the screening visit
* Patients understanding the study, willing to follow the instructions and providing their written Informed Consent Form to participate
* Patients with moderate up severe dry eye with keratoconjunctivitis sicca diagnosed at least 4 weeks before the screening visit
* Patients using artificial tears at least once a day for at least 4 weeks before the screening visit
* Patients with corneal/conjunctival lesions consistent with a diagnosis of keratoconjunctivitis measured by tests of staining: i.e. the overall score of the corneal staining test must be ≥ 3 and ≤ 9 on the 15-point Oxford scale
* And at least one of the following element: Tear volume decreased: must be either present a Schirmer test ≥ 3 mm and ≤ 9 mm / 5 minutes or the sum of 3 consecutive measurements of the tear film break-up time (TBUT) ≤ 30s for at least one eye;
* OSDI score ≥18
* Covered by healthcare insurance.

Exclusion Criteria:

* Patients with medical history of herpetic keratitis, peripheral ulcerative keratitis, sclerites, diabetic retinopathy
* Any systemic disease that is not well controlled for at least 2 months (e.g. lupus, rheumatoid arthritis, thyroiditis…) according to clinical judgment
* Patients using any topical therapies such as non-steroidal anti-inflammatory drugs, cortisone, cyclosporine, vasoconstrictor
* Patients with at least one of the following concomitant ocular inflammatory disease: Stevens Johnson Disease, Atopic Keratoconjunctivitis; Scarlet Eye Pemphigoid
* Patients with anomalies of the eyelid, sucking, infectious conjunctivitis, pterygia, and/or a glaucoma treated with eyedrops
* Presence of graft versus host disease (GVHD)
* Patients who have undergone surgery in the eye, within three months before the study enrolment
* Patients who have undergone corneal transplantation or refractive surgery or plan to undergo any eye surgery in the next four months
* Patients with known or suspected eye allergy
* Patients with a condition or history that, in the opinion of the investigator, may interfere significantly with the subject's participation in the study
* Female pregnant, planning a pregnancy during the study period and nursing an infant
* Patients who are participating or have participated in other clinical trial with investigational drug or device within 30 days prior to screening
* Patients unable to be compliant with the study procedures and requirements, according to the opinion of the investigator
* Patient deprived of liberty by a judicial or administrative decision, or who is under a measure of legal protection (e.g. guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Primary endpoint/clinical performance by Oxford scale | between Day 1 and Day 35 ±4.
  Clinical performance of the medical device under investigation: the between-group comparison of the average variation of the global fluorescein corneal and lissamine green conjunctival staining using the Oxford scale (0 to 15). This refers to the average variation between both time points of the Global Ocular Staining Score of the study eye (GOSS).
  0-5 cornea; 0-5 temporal conjuctiva; 0-5 nasal conjunctiva. Max total score: 15

SECONDARY OUTCOMES:
Secondary endpoint/clinical performance by TBUT test | between Day 1 and Day 35 ±4 and Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of the time obtained at the tear break up time test (TBUT). This full procedure will be performed 3 times per eye and per time point. Each obtained time will be recorded by the investigator in the eCRF. At screening and at baseline visits, the sum of these 3 times for at least one eye to be eligible must be ≤ 30 seconds.
  Conventionally TBUT's measures shorter than 10 seconds can be referred to tear film instability and measures shorter than 5 seconds, usually, are undoubtable sign of dry eye. The longer it takes, the more stable the tear film. A short TBUT is a sign of poor tear film. A positive number change from baseline indicates an increase in TBUT (improvement) and a negative number change from baseline indicates a decrease in TBUT (worsening).
Secondary endpoint/patient reported outcome by DEQS questionnaire | between Day 1 and Day 35 ±4 and Day 1 and Day 84 ±7
  The between-group comparisons of the average variation of Dry Eye-Related Quality-of-Life (DEQS) general score. It is a validated 15-item scale divided into 2 subscales related to dry eye symptoms and its influence on daily life:
  The frequency is scored on a 5-point Likert scale ranging from 0 (no symptom) to 4 (highest frequency).
  • The degree is scored on a 4-point Likert scale ranging from 1 to 4, a larger number indicates a greater burden.
  The summary score ranges from 0 to 100, higher score indicates higher disability. .
Secondary endpoint/safety | between Day 1 and Day 84 ±7
  The description of all adverse events, related and unrelated to the medical devices, anticipated or unanticipated
Secondary endpoint/clinical performance by Oxford scale | between Day 1 and Day 84 ±7
  The between-group comparison of the average variation of the global fluorescein corneal and lissamine green conjunctival staining using the Oxford scale (0-15).This refers to the average variation between both time points of the of the Global Ocular Staining Score of the study eye (GOSS) and the comparison between both treatment groups. -5 cornea; 0-5 temporal conjuctiva; 0-5 nasal conjunctiva. Max total score: 15
Secondary endpoint/clinical performance by Schirmer test | between [Day 1 and Day 84 ±7]
  The between-group comparisons of the average variation of the paper length obtained at the Schirmer Test. The Schirmer test without anesthesia will be here performed to measure the rate of secretion of tears produced by the study eye over 5 minutes.The cut-off value for a severe dry eye in the first one is 6 mm. But the cut-off that will here use will be 9 mm with the following interpretation:
  * Normal = ≥ 10 millimeters (mm) of tears,
  * Dry Eye = ≤ 9 mm of tears A positive number change from baseline indicates an increase in tears (improvement) and a negative number change from baseline indicates a decrease in tears (worsening).
Secondary endpoint/patient reported outcome by OSDI score | between [Day 1 and Day 35 ±4] and [Day 1 and Day 84 ±7]
  The between-group comparisons of the average variation of Ocular Symptoms Disease Index (OSDI) score. The patient's dry eye symptoms will be assessed with the Ocular Surface Disease Index (OSDI). It is a validated 12-questions scale for patients that covers a broad spectrum of ocular surface symptoms, the severity of such symptoms for patients and how these symptoms affect/impact visual function over a 1-week recall period. Its scores range from 0 to 100, with higher scores indicating greater severity of disease.Positive result is considered when the OSDI score is ≥ 18.To be consistent with the IMD indication, patient with moderate to severe dry eye thus with an OSDI ≥ 18 will be selected. If the patient's OSDI score will be strictly below 18 at the screening or baseline visit, s/he will be considered as a screening failure.
  Each item response will be collected in the study database since given separately to patients.

OTHER OUTCOMES:
Investigator's overall treatment satisfaction (PRO) | at [Day 35±4 and Day 84 ±7].
  The between group comparison using on a four-point scale assessing investigator's overall satisfaction on the treatment's clinical performance
  • The between group comparison using on a four-point scale assessing investigator's overall satisfaction on the treatment's clinical performance at [Day 35±4 and Day 84 ±7].
  Overall investigator' satisfaction of the product's clinical performance will be assessed at the end of the patient follow-up period on a four-point scale from 0: very satisfactory, 1: satisfactory; 2: somewhat unsatisfactory; 3: unsatisfactory Safety • The description of all adverse events, related and unrelated to the medical devices, anticipated or unanticipated.
  Exploratory endpoints
  • PROs: the between-group comparisons of the average variation of the DEQS subscale scores between [Day 1 and Day 35 ±4] and [Day 1 and Day 84 ±7].

CONTACTS AND LOCATIONS:
Overall Officials: Marc Labetoulle, MD; Pr, Principal Investigator — CHU KREMLIN-BICETRE
Locations (11):
- France (10):
  - CHU d'Amiens, Amiens
  - Centre Rétine Anjou, Angers
  - Cabinet d'ophtalmologie Fosh, Bordeaux
  - Hopital Saint Vincent de Paul, Lille
  - Hopital Edouard Herriot, Lyon
  - Hôpital Saint Joseph, Marseille
  - Chu Kremlin-Bicetre, Paris
  - APHP - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - CHU Strasbourg, Strasbourg
- Hospital Universitario Miguel Servet, Zaragoza, Spain